CLINICAL TRIAL: NCT00182130
Title: Quality Initiative in Rectal Cancer (QIRC) Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Organization: McMaster University (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: MCT-50013
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Last update posted 2005-09-16 (Estimated); Status verified 2005-07

CONDITIONS: Rectal Cancer
Keywords: rectal cancer; surgery; physician behaviour; knowledge translation
MeSH Terms: conditions — Rectal Neoplasms

INTERVENTIONS:
Procedure: Quality Initiative in Rectal Cancer (QIRC) strategy

SUMMARY:
The Quality initiative in rectal cancer (QIRC) trial will test if a strategy designed to positively influence surgeon practice can decrease hospital rates of permanent colostomy and local tumour recurrence for surgically treated rectal cancer patients.

DETAILED DESCRIPTION:
Approximately 5000 Canadians are annually diagnosed with rectal cancer. For patients undergoing rectal cancer surgery two unfortunate outcomes are permanent colostomy and local tumor recurrence. Research demonstrates that in Ontario, Canada and other parts of the world the standard of care for rectal cancer surgery leaves room for improvement.

This is a multi-center trial that will test if a set of interventions designed to positively influence surgeon practice, titled the Quality Initiative in Rectal Cancer (QIRC) strategy, can improve rates of permanent colostomy and local tumour recurrence for surgically treated rectal cancer patients. Secondary outcomes to be assessed include sexual, bowel, and bladder function, and quality of life. The QIRC strategy consists of a workshop to discuss quality issues in rectal cancer, operative demonstration to demonstrate optimal surgical techniques, the use of opinion leaders, and a postoperative questionnaire designed to prompt surgeons to re-examine their key operative steps. The QIRC strategy is largely designed to teach total mesorectal excision, a new gold standard for rectal cancer surgery that has been shown in non-randomized studies to lower patient rates of permanent colostomy and local tumour recurrence.

Sixteen hospitals across the province of Ontario were allocated by cluster randomization to the QIRC strategy (experimental arm) versus minimal intervention (control arm). All hospitals are high-volume centres - an annual rectal cancer procedure volume of 15 or greater. Hospitals in the control arm represent the normal practice environment. Approximately 700 patients will be assessed. In addition to measuring rates of permanent colostomy and local recurrence of tumour, the study will examine bowel, bladder and sexual function, and overall quality of life among patients.

A positive trial - better results in hospitals that receive the intervention - may suggest that to effectively influence surgeon practice, resource intense approaches are necessary along with active buy-in from the surgical community.

ELIGIBILITY:
Inclusion Criteria:

Hospital inclusion criteria:

1. An Ontario hospital with a procedure volume of 15 or more major rectal cancer resections per year for fiscal years 1996 to 1998.

Patient inclusion criteria:

1. Consecutive patients at each participating site who underwent major rectal cancer surgery.
2. Tumor located within 15 cm of anal verge by rigid sigmoidoscopy, or, at or below the level of the sacral promontory at the time of surgery.

Exclusion Criteria:

-

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 691
Dates: Start 2002-05; Study Completion 2007-06

PRIMARY OUTCOMES:
Hospital rate of permanent colostomy
Hospital rate of local recurrence

SECONDARY OUTCOMES:
Bowel, bladder and sexual function
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Marko Simunovic, MD, Principal Investigator — McMaster University

REFERENCES:
- [Derived] Simunovic M, Coates A, Goldsmith CH, Thabane L, Reeson D, Smith A, McLeod RS, DeNardi F, Whelan TJ, Levine MN. The cluster-randomized Quality Initiative in Rectal Cancer trial: evaluating a quality-improvement strategy in surgery. CMAJ. 2010 Sep 7;182(12):1301-6. doi: 10.1503/cmaj.091883. Epub 2010 Aug 9. PMID 20696797